CLINICAL TRIAL: NCT01782430
Title: PREoxygenation for the Intubation of Hypoxemic Patients: Comparison of Standard Oxygenation, High Flow Nasal Oxygen Therapy, and NonInvasive Ventilation
Acronym: PREONIV
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Hopital Gabriel Montpied (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0141; 2012-A00778-35 (Registry Identifier: 2012-A00778-35)
Record Dates: First submitted 2013-01-31; First posted 2013-02-01 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Adult Patients; Requiring Intubation; Hypoxemia (Defined by PaO2/FiO2( Fraction of Inspired Oxygen) Below 200); Patient Covered by French Health Care System
Keywords: Preoxygenation; Intubation
MeSH Terms: conditions — Hypoxia

ARMS (3):
- Standard oxygenation (Experimental): Prospective randomized clinical multicentric study in ICU, comparing standard oxygenation, high flow nasal oxygen therapy and non invasive ventilation (NIV) , with pulse oxymetry values (SpO2), during preoxygenation for hypoxemic patients
  Interventions: Procedure: - standard oxygenation
- High flow nasal oxygen therapy (Experimental): Prospective randomized clinical multicentric study in ICU, comparing standard oxygenation, high flow nasal oxygen therapy and non invasive ventilation (NIV) , with pulse oxymetry values (SpO2), during preoxygenation for hypoxemic patients
  Interventions: Procedure: - standard oxygenation
- invasive ventilation (VNI) (Other): Prospective randomized clinical multicentric study in ICU, comparing standard oxygenation, high flow nasal oxygen therapy and non invasive ventilation (NIV) , with pulse oxymetry values (SpO2), during preoxygenation for hypoxemic patients
  Interventions: Procedure: - standard oxygenation

INTERVENTIONS:
Procedure: - standard oxygenation

SUMMARY:
Prospective, randomized clinical multicentric study, in ICU, during preoxygenation for the intubation of hypoxemic patients.

DETAILED DESCRIPTION:
Prospective randomized clinical multicentric study in ICU, comparing standard oxygenation, high flow nasal oxygen therapy and non invasive ventilation (NIV) , with pulse oxymetry values (SpO2), during preoxygenation for hypoxemic patients

ELIGIBILITY:
Inclusion Criteria:

* adults patients
* requiring intubation and hypoxemia (defined by PaO2/FiO2 below 200)
* patient covered by french health care system

Exclusion Criteria:

* patient refusal
* intubation for other causes (excluding hypoxemia)
* impossibility to measure pulse oxymetry value
* contraindication for NIV : vomiting
* NIV intolerance
* cardiac arrest during intubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
least pulse oxymetry value | at day 1

SECONDARY OUTCOMES:
pulse oxymetry value (at the end of preoxygenation) | at 5 minutes and at 30 minutes after intubation
Partial pressure of arterial oxygen (PaO2) | at day 1
Regurgitation rate | at day 1
oxyhemoglobin desaturation below 80 % | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien PERBET, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France